CLINICAL TRIAL: NCT03947554
Title: Study of the Efficacy of Panax Ginseng Herbal Preparation HRG80 for Prevention and Mitigation of the Symptoms of Stress in Healthy Subjects
Brief Title: Ginseng HRG80 in Stress and Fatigue
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EuroPharma, Inc. (Industry)
Collaborators: Botalys SA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EP-1005
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-05

CONDITIONS: Psychological Stress
Keywords: Panax ginseng; Red ginseng; Korean ginseng; Adaptogen
MeSH Terms: conditions — Stress, Psychological | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HRG80 Panax ginseng (Experimental): Panax ginseng standardized to 63.4 mg of total ginsenosides taken orally once daily in the morning after a meal.
  Interventions: Dietary Supplement: HRG80 Panax ginseng
- Panax ginseng (Active Comparator): Panax ginseng standardized to 19.6 mg of total ginsenosides taken orally once daily in the morning after a meal.
  Interventions: Dietary Supplement: Panax ginseng
- Placebo (Placebo Comparator): Placebo capsule containing brown sugar and rice flour, taken orally once daily in the morning after a meal.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HRG80 Panax ginseng — Panax ginseng containing 63.4 mg ginsenosides
  Arms: HRG80 Panax ginseng
Dietary Supplement: Panax ginseng — Panax ginseng containing 19.6 mg ginsenosides
  Arms: Panax ginseng
Dietary Supplement: Placebo — 800 mg excipient
  Arms: Placebo

SUMMARY:
This study evaluates the effects of a specific herbal preparation of Panax ginseng in preventing symptoms of stress in healthy individuals.

DETAILED DESCRIPTION:
HRG80 is an herbal preparation of Panax ginseng with a higher concentration of bioavailable ginsenosides than typical Korean ginseng. This study will test whether HRG80 is effective at preventing symptoms of stress, such as fatigue, impaired memory, difficulty in concentration, attention deficit, restlessness, and irritation related to daily work situations of healthy individuals in comparison to placebo and a standard Pananx ginseng with a lower concentration of ginsenosides.

ELIGIBILITY:
Inclusion Criteria:

* Individuals experiencing at least one symptom of stress and fatigue during 8 hours of mental work with a computer.
* Men and women ages 18-65 (all races and ethnicities)
* Able to understand and participate in an 11-week study

Exclusion Criteria:

* Taking medicine or dietary supplements which may have potential effects on cognitive function
* Consuming more than 1 cup of coffee daily (in the morning).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale (PSS) from baseline to the last day of treatment | Two weeks
  The Perceived Stress Scale is a psychological instrument for measuring the perception of stress by an individual. Scores from 0-13 indicate low stress, 14-26 is considered moderate stress, and scores from 27-40 indicate high perceived stress. The primary outcome is the change in the baseline PSS score for HRG80 versus standard Panax ginseng and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Areg Hovhannisyan, PhD, Dr Sci, Principal Investigator — Sports Medicine and Anti-Doping Service Republican Centre
Locations (1):
- Sports Medicine and Anti-Doping Service Republican Centre, Yerevan, Armenia